CLINICAL TRIAL: NCT06193486
Title: A Phase I Clinical Trial of an Infusion of Autologous Gamma Delta T Cells Genetically Engineered With a Chimeric Receptor to Target the Prostate Stem Cell Antigen in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Autologous Gamma Delta T Cells to Target Prostate Stem Cell Antigen in mCRPC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22344
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Participants will undergo leukapheresis followed by lymphodepletion and infusion of MSGV1-PSCA-8T28Z. The lymphodepletion regimen includes cyclophosphamide (500 mg/m2) and fludarabine (30 mg/m2) administered over 3 days (Days -5, -4, -3). The standard "3+3" design will be used to guide dose escalation/de-escalation decisions based on the cumulative number of patients who experience a dose limiting toxicity (DLT) at the current dose. The first cohort of 3 patients will be treated at dose level 1.
  The target maximum doses infused at each dose level is:
  Dose Level 1: 1x10^5 cells/kg Dose Level 2: 3x10^5 cells/kg Dose Level 3: 1x10^6 cells/kg Dose Level 4: 3x10^6 cells/kg Dose Level 5: 1x10^6 cells/kg
  Interventions: Biological: MSGV1-PSCA-8T28Z; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Expansion (Experimental): Participants will undergo leukapheresis followed by lymphodepletion and infusion of MSGV1-PSCA-8T28Z. Lymphodepletion will include 3 days of treatment with fludarabine (30 mg/m^2) and cyclophosphamide (500 mg/m^2) prior to study day 0. Participants will then receive MSGV1-PSCA-8T28Z at the dose level determined to be the Maximum Tolerated Dose (MTD) in the dose escalation portion of the study.
  Interventions: Biological: MSGV1-PSCA-8T28Z; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: MSGV1-PSCA-8T28Z — Autologous Gamma Delta T Cells Genetically Engineered with a Chimeric Receptor to Target the Prostate Stem Cell Antigen.
Drug: Fludarabine — Fludarabine is an antimetabolite given prior to lymphodepletion.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide is a nitrogen mustard-derivative, polyfunctional alkylating agent given prior to lymphodepletion.

SUMMARY:
This is a phase 1 single center clinical trial for patients with end stage Metastatic Castration Resistant Prostate Cancer who have progressed through standard of care treatment options and are on zoledronate for bone metastases. This clinical trial includes a dose-escalation phase and dose-expansion phase to assess the safety and preliminary efficacy of treatment with autologous T cells genetically modified to express Prostate stem cell antigen.

ELIGIBILITY:
Inclusion Criteria:

* Men with metastatic castration-resistant prostate cancer (CRPC) to the bone with evidence of imaging progression based on the PCWG3 criteria.
* Prior therapies with at least one line of chemotherapy and one new androgen receptor targeted therapy (abiraterone, enzalutamide, apalutamide, or darolutamide).
* For patients who are on zoledronic acid a booster dose of zoledronic acid is required if the last dose of zoledronic acid is >4 weeks prior to lymphodepletion chemo. If a patient is receiving denosumab, the next dose of denosumab needs to be changed to zoledronic acid and he needs to receive at least 1 dose of zoledronic acid prior to lymphodepletion chemotherapy. If a patient is not on zoledronic acid or denosumab, he needs to receive at least 2 doses of every 4 weeks of zoledronic acid prior to lymphodepletion chemotherapy. Zoledronic acid is recommended not to be resumed prior to week 8. After week 8, the resumption of zoledronic acid and the subsequent zoledronic acid treatment will be at the discretion of the treating physician.
* No anticancer therapy (chemotherapy, biologic therapy, radiation or immunotherapy) in the 3 weeks before the T cell infusion (and all hematologic effects have resolved). No prior treatment with Radium 223 or Puvicto within 3 months of T cell infusion. No prior immunotherapy with checkpoint blockade (e.g., PD-1 inhibitor, PDL1 inhibitor, or CTL4- antagonist or similar agent) in the 6 months before the T cell infusion (and all clinically significant related side effects must be resolved).
* Males age 18 years or older.
* ECOG performance status less than or equal to 2 (or Karnofsky Performance Status greater than or equal to 70%).
* Participants must have adequate organ and marrow function as defined by the protocol.
* Life expectancy of at least 6 months.
* The effects of CAR T cell infusion on the developing human fetus are unknown. Although patients who are eligible for this study will not have childbearing potential, any patient the treating doctor or investigator deems to have child fathering potential must agree to use adequate contraception from the time of screening to at least 6 months after administration of gamma delta enriched T cell infusion. Any female partner(s) with childbearing potential, of these participants, should also use adequate contraception during the same time period.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known active hepatitis B infection, known history of hepatitis C or HIV infection.
* Known dental issues like osteonecrosis of jaw that excludes the use of zoledronic acid
* Any of the following cardiac conditions: Clinically significant heart disease (New York Heart Association class 3 or 4) or symptomatic congestive heart failure, Myocardial infarction less than 6 months before enrollment, History of clinically significant ventricular arrhythmia or unexplained syncope that is not believed to be vasovagal in nature or due to dehydration, History of severe non-ischemic cardiomyopathy with ejection fraction less than 20%, or Findings on baseline ECG or ECHO that, in the opinion of the patient's treating physician or investigator, would require medical intervention before anticancer therapy
* Active autoimmune disease (excluding autoimmune thyroid disease on a stable thyroid regimen). Such conditions include but are not limited to systemic lupus erythematous, rheumatoid arthritis, ulcerative colitis, Crohn's disease, and temporal arteritis.
* Known or suspected leptomeningeal disease and patients with metastases to the brain stem, midbrain, pons, or medulla.
* Known or suspected untreated brain metastases. Patients with radiographically stable, asymptomatic previously irradiated lesions are eligible provided patient is greater than 4 weeks beyond completion of cranial irradiation and greater than 3 weeks off of corticosteroid therapy at the time of study intervention.
* Prior history of clinically significant seizure disorder (e.g., not including childhood febrile seizures).
* Any concurrent active malignancies, defined as malignancies requiring any therapy other than expectant observation, because adverse events (AEs) resulting from these malignancies, or their treatment may confound our assessment of the safety of adoptive T cell therapy for ovarian cancer.
* Any of the following within 28 days of first date of study treatment: Serious uncontrolled medical illness or disorder that in the opinion of the treating physician would make the patient ineligible for the study, or Active uncontrolled infection (with the exception of uncomplicated urinary tract infection)
* Prior history of pancreatitis.
* Any other issue which, in the opinion of the treating physician or principal investigator, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2029-01-13 (Estimated); Study Completion 2033-12-13 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MSGV1-PSCA-8T28Z | Up to 30 days post transplant
  MTD of MSGV1-PSCA-8T28Z based on Dose Limiting Toxicity (DLT) in patients with Metastatic Castration-Resistant Prostate Cancer.

SECONDARY OUTCOMES:
Best Prostate Specific Antigen (PSA) Response rate | Up to 5 years
  Best PSA Response rate, which will be measured by percentage of patients who had 50% decline in PSA.
Radiographic progression-free survival (rPFS) | Up to 5 years
  rPFS is defined as the duration of time from start of treatment to time of progression or death.
Percentage of circulating tumor cell count conversion from above 5/ml to below 5/ml. | Up to 5 years
  The Circulating tumor cell conversion rate from above 5 to less than 5 will be used as a response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, PhD, Principal Investigator — Moffitt Cancer Center; Daniel Abate-Daga, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided